CLINICAL TRIAL: NCT06955169
Title: MOMENTUM-1: A Multicenter, Randomized, Open-Label, Phase II Study of [177LU]LU-DOTATATE in Adults With Progressive Intracranial Grade 1-3 Meningioma
Brief Title: Comparing the Radiopharmaceutical Drug, [177Lu]Lu-DOTATATE, to Standard of Care Treatment for Patients With Meningioma That Has Come Back After Prior Treatment
Acronym: MOMENTUM-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RTOG Foundation, Inc. (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 3523; CAAA601A1US13R (Other: Novartis Pharmaceuticals, Inc.)
Record Dates: First submitted 2025-04-22; First posted 2025-05-02 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Meningioma
Keywords: MOMENTUM-1; Meningioma; Advanced Intracranial Meningioma; SSTR2; Radiopharmaceuticals; Theranostics; Radioligand Therapy; Lu-DOTATATE; Lutathera
MeSH Terms: conditions — Meningioma | interventions — lutetium Lu 177 dotatate; Bevacizumab; Everolimus; Hydroxyurea; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- [177Lu]Lu-DOTATATE (Experimental): Study participants receive [177Lu]Lu-DOTATATE
  Interventions: Drug: [177Lu]Lu-DOTATATE
- Control (Other): Study participants receive Local Standard of Care (SOC) Therapy. Control Arm participants crossover to [177Lu]Lu-DOTATATE at progression
  Interventions: Other: Standard of Care treatments

INTERVENTIONS:
Drug: [177Lu]Lu-DOTATATE — The treatment regimen consists of 4 (+2 optional) administrations of [177Lu]Lu-DOTATATE. The recommended interval between infusions is 4 weeks (+ 7 days).
  Other Names: Lutathera
  Arms: [177Lu]Lu-DOTATATE
Other: Standard of Care treatments — Treatments will occur at the discretion and based on clinical judgement of the local and treating investigator. Local SOC therapy with one of the following agents: bevacizumab, everolimus, hydroxyurea, or sunitinib.
  Other Names: Avastin (bevacizumab), Afinitor (everolimus), Hydrea (hydroxyurea), Hydroxycarbamide (hydroxyurea), Sutent (sunitinib)
  Arms: Control

SUMMARY:
This is an open-label, multicenter, randomized, phase 2 clinical study to evaluate the efficacy of [177Lu]Lu-DOTATATE in patients with progressive grade 1-3 intracranial meningioma.

DETAILED DESCRIPTION:
Study participants will be randomized by a 2:1 ratio to receive either [177Lu]Lu-DOTATATE or standard of care therapy as deemed appropriate by the local investigator. At time of progression, participants on the standard of care arm may cross-over to the [177Lu]Lu-DOTATATE alternative treatment arm.

ELIGIBILITY:
Inclusion Criteria:

STEP 1 REGISTRATION

* Aged >= 18 years
* Histologically confirmed diagnosis of WHO grade 1-3 meningioma
* Presence of measurable contrast-enhancing disease on gadolinium-enhanced MRI brain scan defined as at least one lesion with two perpendicular diameters measuring ≥10 mm on two or more axial slices (≤ 5 mm interslice thickness, ≤ 1 mm interslice gap) per current RANO meningioma criteria
* Progression of disease determined by local radiology review per current RANO meningioma criteria, defined as

  * ≥ 15% increase in sum of product of perpendicular measurements of up to 5 measurable target lesions within the last 6 months, or
  * ≥ 25% increase in sum of product of perpendicular measurements of up to 5 measurable target lesions within the last 12 months, or
  * Development of a new measurable lesion
* The following scans must be available for submission for central radiology review:

  * Pre-progression gadolinium-enhanced MRI brain scan
  * Progression gadolinium-enhanced MRI brain scan

STEP 2 REGISTRATION

* Progression of disease determined by central radiology review per current RANO meningioma criteria, defined as

  * ≥ 15% increase in sum of product of perpendicular measurements of up to 5 measurable target lesions within the last 6 months, or
  * ≥ 25% increase in sum of product of perpendicular measurements of up to 5 measurable target lesions within the last 12 months, or
  * Development of a new measurable lesion.
* [68Ga]Ga-DOTATATE uptake on PET-CT. Positive uptake is defined as uptake at least as high as liver, based on the uptake in at least one target lesion.
* If randomized to the control (standard of care) arm, both the patient and investigator must agree NOT to receive SSTR2-targeted therapy, surgical resection, or radiation therapy.
* Patients must be willing and able to undergo regular MRI scans of the brain and [68Ga]Ga-DOTATATE PET-CT imaging during the study.
* Patients must have recovered to CTCAE grade ≤1 or pretreatment baseline from clinically significant adverse events related to prior therapy (exclusions include alopecia, lymphopenia, sensory neuropathy ≤ grade 2, or other ≤ grade 2 not constituting a safety risk based on the investigator's judgment).
* Adequate organ and bone marrow function as defined below (within 28 days prior to step 2 registration):

  * Absolute neutrophil count (ANC) ≥ 1500/mm3
  * Platelet count ≥ 75,000/mm3
  * Hemoglobin ≥ 8 g/dL
  * Creatinine clearance (calculated by the Cockroft-Gault method) ≥40mL/min
  * Total serum bilirubin ≤ 3 x ULN (except participants with Gilbert's Syndrome, who can have a total bilirubin ≤ 5 x ULN)
  * Potassium within normal limits.

Exclusion Criteria:

* Patients with a clinical diagnosis of NF2-related schwannomatosis or with a known molecular diagnosis of NF2-related schwannomatosis.
* Patients with radiation-associated meningiomas.
* Patients with known intraspinal meningiomas or meningioma metastases outside the skull/spinal column.
* Prior SSTR2-targeted therapy, e.g. Somatostatin LAR or short-acting Octreotide.
* Unstable neurological symptoms requiring steroids to control symptoms at a dose of >2 mg of dexamethasone (or equivalent) daily within 28 days prior to step 2 registration.
* Patients requiring immediate local therapy (e.g. surgical resection).
* Surgical procedure within the timeframes listed below, prior to step 2 registration.

  * 28 days from any prior craniotomy
  * 7 days from stereotactic biopsy Note: There is no limit to the number of prior surgical interventions
* Treatment within the timeframes specified below, prior to step 2 registration.

  * 28 days (or 5 half-lives, whichever is longer) for cytotoxic chemotherapy, biologic agent, investigational agent or any other systemic agent prescribed for the purpose of treating meningioma
  * 6 weeks from nitrosoureas Note: There is no limit to the number of prior systemically administered therapeutic agents.
* Prior external beam radiation, interstitial brachytherapy or stereotactic radiosurgery cumulative radiation dose of > 70 Gy or the last dose of radiotherapy < 24 weeks (6 months) prior to step 2 registration
* Peptide receptor radionuclide therapy at any time prior to registration.
* Known hypersensitivity to somatostatin analogues or any component of the [68Ga]Ga- DOTATATE or [177Lu]Lu-DOTATATE formulations.
* Active infection requiring current use of intravenous therapy with antibiotics.
* Active cardiovascular disease: cerebral vascular accident/stroke (≤ 6 months prior to registration), myocardial infarction (≤ 6 months prior to registration), congestive heart failure (≥ NYHA class II), unstable angina pectoris, or serious cardiac arrhythmia requiring medication.
* An active malignancy ≤ 3 years. Note: Patients with a malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Pregnant and/or breastfeeding patients who are unwilling to discontinue breast feeding.
* Participants of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2030-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Assessed up to 4 years
  PFS defined as the time from randomization to date of disease progression per current RANO meningioma criteria or death, whichever occurs first

SECONDARY OUTCOMES:
Progression free survival at 6 months (PFS-6) | 6 months
  Proportion of participants alive without progression at 6 months assessed per RANO meningioma criteria
Overall Survival at 12 months (OS-12) | 12 months
  Proportion of participants alive at 12 months
Overall survival (OS) | Assessed up to 4 years
  Time from randomization to death from any cause
Progression-free Survival after cross-over (PFS2) | Assessed up to 4 years
  Time from cross-over to disease progression per RANO meningioma criteria or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | Assessed up to 4 years
  Proportion of patients achieving complete response, partial response, minor response or stable disease as per RANO meningioma criteria
Objective response rate (ORR) | Assessed up to 4 years
  Proportion of patients achieving complete or partial response as per RANO meningioma criteria.
Number of participants by highest grade treatment-emergent adverse event (TEAE): | Assessed up to 4 years
  Number of participants experiencing the highest grade TEAE, graded according to CTCAE version 5.0 (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life-threatening, Grade 5 = death related to adverse event).
Number of participants who discontinue treatment due to TEAE | Assessed up to 4 years
  Number of participants who discontinue treatment as a result of treatment-emergent adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Erik P Sulman, MD,PhD, Principal Investigator — NYU Langone Health; Sylvia C Kurz, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Piedmont Healthcare, Atlanta, Georgia, United States